CLINICAL TRIAL: NCT01284413
Title: Phase I/II Study of Gemcitabine/Cisplatin/S-1(GCS) Combination Therapy for Patients With Advanced Biliary Tract Cancer
Brief Title: Gemcitabine/Cisplatin/S-1(GCS) Combination Therapy for Patients With Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1002; UMIN000004468 (Registry Identifier: UMIN)
Record Dates: First submitted 2011-01-03; First posted 2011-01-27 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — S 1 (combination); Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1, Gemcitabine, Cisplatin (Experimental)
  Interventions: Drug: S-1, Gemcitabine, Cisplatin

INTERVENTIONS:
Drug: S-1, Gemcitabine, Cisplatin — S-1 is given daily for 7 consecutive days and gemcitabine and cisplatin are infused on day1. The cycle is repeated every 2 weeks.
  Other Names: S-1;TS-1, Gemcitabine;gemzer, Cisplatin;Cispulan

SUMMARY:
The objective of this study is to evaluate the safety of GCS therapy for phase I and efficacy of GCS therapy for phase II.

DETAILED DESCRIPTION:
Biliary tract cancer is one of the most lethal malignancies worldwide, with surgery representing the only potentially curative treatment for this disease. However, many patients are diagnosed too late for curative resection, and even if surgery can be performed, the likelihood of relapse is very high. Over the past decade, gemcitabine has been widely used to treat unresectable or recurrent biliary tract cancer patients. In the ABC-02 study, the first prospective multicenter phase III study in this field, gemcitabine/cisplatin combination chemotherapy was compared with gemcitabine monotherapy and found that the combination regimen significantly prolonged MST (from 8.1 to 11.7 months; P < 0.001). Gemcitabine/cisplatin combination therapy is now considered to be the standard regimen for advanced biliary tract cancer. S-1 is an oral fluoropyrimidine prodrug that has confirmed efficacy against various solid tumors, both alone and in combination with other cytotoxic drugs. S-1 monotherapy has yielded good results against advanced biliary tract cancer and gemcitabine/S-1 combination therapy has yielded promising results with acceptable toxicity levels for patients with advanced biliary tract cancer. In this study, we aimed to determine the safety and efficacy of adding S-1 to gemcitabine/cisplatin combination regimen for advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with cytologically or histologically proved biliary tract cancer 2. age >=20 years 3. PS 0-2 4. No prior history of chemotherapy or radiotherapy. Patients who have undergone adjuvant chemotherapy are eligible if at least 6 months have passed since the last administration.

  5. Adequate bone marrow function (neutrophil count >=1,500/mm3, and platelet count >=100,000/mm3), liver function (total bilirubin >=3 mg/dL and AST/ALT >=150 IU/L), and renal function (creatinine clearance >=60 mL/min) 6.No other serious comorbid disease 7.Adequate oral intake 8.Provided written informed consent

Exclusion Criteria:

* 1. Patients with interstitial pneumonia or pulmonary fibrosis 2. Patients with uncontrollable diabetes mellitus, liver disease, angina pectoris or a new onset of myocardial infarction within 3 months 3. Patients with severe active infection 4. Patients who are pregnant or lactating, or have an intention to get pregnant 5. Patients with a history of severe drug allergy 6. Patients with other serious comorbid disease 7. Patients with mental disease 8. Patients who are judged inappropriate for the entry into the study by the principle doctor 9. Patients with watery diarrhea

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
one year survival rate | 2 years
  The primary endpoint is designated to evaluate overall survival rate at 12-month. Secondary endpoints include response rate according to RECIST 1.1 and the incidence of adverse events evaluated by CTCAE v 4.0.

SECONDARY OUTCOMES:
Toxicity and response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Etsuro Hatano, MD, PhD, Study Director — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Kanai M, Hatano E, Kobayashi S, Fujiwara Y, Marubashi S, Miyamoto A, Shiomi H, Kubo S, Ikuta S, Yanagimoto H, Terajima H, Ikoma H, Sakai D, Kodama Y, Seo S, Morita S, Ajiki T, Nagano H, Ioka T. A multi-institution phase II study of gemcitabine/cisplatin/S-1 (GCS) combination chemotherapy for patients with advanced biliary tract cancer (KHBO 1002). Cancer Chemother Pharmacol. 2015 Feb;75(2):293-300. doi: 10.1007/s00280-014-2648-9. Epub 2014 Dec 5. PMID 25477010